CLINICAL TRIAL: NCT04317053
Title: Multi-Center Randomized Controlled Trial of Relay- NYC's Nonfatal Overdose Response Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-01547
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Site-Directed Care (SDC) (No Intervention): Site-specific existing interventions delivered to patients with OUD as part of ED care. At a minimum SDC arm patients will receive from the study research team OD education and naloxone distribution (OEND), a list of opioid treatment programs, and an informational flyer about Relay.
- Relay program (peer navigation) (Experimental): Relay is a novel program that engages and intervenes with individuals in the ED following an opioid OD and for the next 90 days, with the goal of preventing subsequent OD events. Relay is delivered by trained peer navigators, who are DOHMH staff with lived substance use experience. Relay navigators provide counseling, linkage to services, and OD prevention education.
  Interventions: Behavioral: RELAY

INTERVENTIONS:
Behavioral: RELAY — Relay is a novel program that engages and intervenes with individuals in the ED following an opioid OD and for the next 90 days, with the goal of preventing subsequent OD events. Relay is delivered by trained peer navigators, who are DOHMH staff with lived substance use experience. Relay navigators provide counseling, linkage to services, and OD prevention education.
  Arms: Relay program (peer navigation)

SUMMARY:
The New York City (NYC) Department of Health and Mental Hygiene (DOHMH) has implemented Relay, a novel program that engages and intervenes with individuals in the ED following an opioid OD and for the next 90 days, with the goal of preventing subsequent OD events. The proposed randomized controlled trial will evaluate the impact of Relay on preventing subsequent opioid-related adverse events. A total of 350 eligible individuals with nonfatal opioid OD presenting to one of four participating EDs will be enrolled and randomized to one of two arms: 1) site-directed care (SDC) or 2) Relay-peer-delivered OD education and treatment linkage, including 90 days of peer navigation. Outcomes will be measured for 12 months through interviews and administrative health data.

DETAILED DESCRIPTION:
Relay is a novel program that engages and intervenes with individuals in the ED following an opioid OD and for the next 90 days, with the goal of preventing subsequent OD events. Relay is delivered by trained peer navigators, who are DOHMH staff with lived substance use experience. Relay navigators provide counseling, linkage to services, and OD prevention education.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* English- or Spanish-speaking
* Patient at a participating ED with nonfatal opioid OD.
* Currently residing in NYC

Exclusion Criteria:

* Unable to provide informed consent
* Currently incarcerated, currently living in another controlled environment prohibiting research contacts, or currently in police custody
* Known to be currently pregnant
* Already participating in the study (patients will only be enrolled into the study once)
* Already actively engaged in the Relay program (within the 90-day program window)
* Speaks only Spanish, at a site and time period when no Spanish-speaking RA is available

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Doran, MD, Principal Investigator — New York University
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months following article publication and ending 6 years after any reporting, publication, or presentation.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Upon request, study investigators will provide the research dataset to qualified investigators under a Data Use Agreement (DUA) that will require approval of the study Principal Investigators and each of the primary research team participating agencies (NYU and NYC Department of Health and Mental Hygiene).

REFERENCES:
- [Derived] Doran KM, Welch AE, Kepler KL, Jeffers A, Chambless D, Cowan E, Wittman I, Regina A, Siu K, Bailey VS, Rostam-Abadi Y, Kennedy J, Kunins HV, Gwadz M, Shelley D, Cleland CM, McNeely J. Peer Navigator Intervention and Opioid-Related Adverse Events for Emergency Department Patients: A Randomized Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2555903. doi: 10.1001/jamanetworkopen.2025.55903. PMID 41649817
- [Derived] Doran KM, Welch AE, Jeffers A, Kepler KL, Chambless D, Cowan E, Wittman I, Regina A, Chang TE, Parraga S, Tapia J, Diaz C, Gwadz M, Cleland CM, McNeely J. Study protocol for a multisite randomized controlled trial of a peer navigator intervention for emergency department patients with nonfatal opioid overdose. Contemp Clin Trials. 2023 Mar;126:107111. doi: 10.1016/j.cct.2023.107111. Epub 2023 Feb 4. PMID 36746325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Started | 126 | 127
Completed | 122 | 125
Not Completed | 4 | 2
Not completed — Withdrawn (screen failure) | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation) | Total
Number analyzed (Participants) | 122 | 125 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (14.5) | 48.7 (13.8) | 49.5 (14.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 91 | 99 | 190
  Unknown/Not Reported | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 56 | 126
  Not Hispanic or Latino | 52 | 69 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 37 | 80
  White | 34 | 42 | 76
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 34 | 38 | 72
Region of Enrollment [Number; unit: participants]
  United States | 122 | 125 | 247

OUTCOME MEASURES:

1. Primary Outcome: Number of Opioid-related Adverse Events
Description: Opioid-related adverse events includes fatal and non-fatal opioid-involved overdose as well as substance use-related emergency department (ED) visits. ED visits and fatal overdoses in the 12-month period after baseline will be captured in administrative data sources. Other non-fatal opioid-involved overdose events will be captured by self-report in follow-up interviews through six months after baseline, and estimated for the second half of the 12-month follow-up period.
Time Frame: Up to Month 12
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 122 | 125
Events | 4.15 (9.58) | 3.24 (4.76)

2. Secondary Outcome: Number of Participants Who Initiate Medication for Opioid Use Disorder (MOUD)
Description: MOUD is defined as use of methadone, buprenorphine, or naltrexone that is prescribed by an office-based provider or provided by a treatment program as treatment for OUD. Initiation is defined as receiving MOUD within the 90 days following the index visit, for individuals who received no MOUD for at least 2 weeks prior to the index visit.
Time Frame: Up to Month 3
Population: Not all participants involved in the study completed all outcome measure data collection visits for each individual outcome measure. Thus, not all participants who completed the study are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 97 | 93
Percentage of participants | 14.4 [8.8 to 22.8] | 16.1 [10.0 to 24.9]

3. Secondary Outcome: Overdose Risk Behavior Questionnaire Score
Description: 13-item questionnaire assessing overdose risk behaviors. Items are rated on a Likert scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 52; higher scores indicate more prevalent overdose risk behaviors.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 122 | 125
score on a scale | 8.22 (6.35) | 8.9 (8.13)

4. Secondary Outcome: Overdose Risk Behavior Questionnaire Score
Description: as for outcome 3
Time Frame: Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 62 | 66
score on a scale | 4.39 (6.51) | 6.52 (6.6)

5. Secondary Outcome: Overdose Risk Behavior Questionnaire Score
Description: as for outcome 3
Time Frame: Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 72 | 75
score on a scale | 4.49 (6.61) | 6.6 (7.01)

6. Secondary Outcome: Overdose Risk Behavior Questionnaire Score
Description: as for outcome 3
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 69 | 70
score on a scale | 3.77 (6.14) | 6.46 (8.13)

7. Secondary Outcome: Time to Next Opioid-Involved Overdose
Description: Time to next opioid-involved overdose from the time of baseline, by self-report.
Time Frame: Up to Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 22 | 27
days | 68.0 (49.3) | 57.8 (51.4)

8. Secondary Outcome: Number of Emergency Deparment (ED) Visits for Any Cause
Description: Frequency of ED visits for any cause (including visits that are not substance use-related) will be measured, using administrative data, to assess whether there are differences in overall acute care use representing potentially negative health events.
Time Frame: Up to Month 12
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 122 | 125
Visits | 6.73 (12.9) | 6.28 (8.85)

9. Secondary Outcome: Number of ED Visits for Other (Non-OD) Substance Use Reasons
Description: Frequency of ED visits for other (non-OD) substance use will be measured, using administrative data.
Time Frame: Up to Month 12
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 122 | 125
Visits | 2.98 (8.62) | 2.26 (4.03)

10. Secondary Outcome: Number of Opioid Overdose-Related ED Visits
Description: Frequency of ED visits for opioid overdose will be measured, using administrative data
Time Frame: Up to Month 12
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 122 | 125
Visits | 0.402 (1.28) | 0.376 (0.964)

11. Secondary Outcome: Percentage of Participants Who Self-Report Opioid-Involved Overdose
Description: Includes non-fatal overdose that did or did not result in an ED visit, by self report.
Time Frame: Month 1
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 62 | 66
Percentage of participants | 11.3 | 16.7

12. Secondary Outcome: Percentage of Participants Who Self-Report Opioid-Involved Overdose
Description: Includes non-fatal overdose that did or did not result in an ED visit, by self report.
Time Frame: Month 3
Measure: Number; unit: Percentage of participants
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 74 | 76
Percentage of participants | 24.3 | 31.6

13. Secondary Outcome: Percentage of Participants Who Self-Report Opioid-Involved Overdose
Description: Includes non-fatal overdose that did or did not result in an ED visit, by self report.
Time Frame: Month 6
Measure: Number; unit: Percentage of participants
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
Number analyzed (Participants) | 76 | 74
Percentage of participants | 30.3 | 37.8

ADVERSE EVENTS:
Time Frame: 12 months
Description: All mortality was assessed by the NYC Department of Health and Mental Hygiene by examining vital statistics records for all study participants.
Arm/Group | Site-Directed Care (SDC) | Relay Program (Peer Navigation)
All-Cause Mortality (participants affected / at risk) | 23/122 | 21/125
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/125
Other Adverse Events (participants affected / at risk) | 0/122 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT04317053/Prot_SAP_002.pdf
  • Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04317053/ICF_001.pdf